CLINICAL TRIAL: NCT00844727
Title: Coxib-inhibition of Duodenal Polyp Growth in Familial Adenomatous Polyposis
Brief Title: Coxib-inhibition of Duodenal Polyp Growth in FAP
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Drug withdrawal
Sponsor: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RH01/01
Record Dates: First submitted 2009-02-13; First posted 2009-02-16 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2009-02

CONDITIONS: Duodenal Polyposis
MeSH Terms: interventions — rofecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Rofexocib 25 mg OD, 1 year treatment
  Interventions: Drug: Rofecoxib
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Rofecoxib
  Arms: 1
Drug: placebo — placebo pills
  Arms: 2

SUMMARY:
Preliminary data indicate a protective effect on the development of duodenal polyps by coxib treatment. The hypothesis of the present study is that normal therapy doses of rofecoxib for 1 year would stop or reverse the development of premalignant adenomatous lesions in the duodenal mucosa of FAP patients.

ELIGIBILITY:
Inclusion Criteria:

* FAP patient with previous colectomy and confirmed polyposis

Exclusion Criteria:

* Pregnancy
* Malignancy
* NSAID hypersensitivity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2003-09; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Medicine, Rikshospitalet, Oslo, Oslo County, Norway